CLINICAL TRIAL: NCT05990309
Title: ASSESSMENT OF TRISTETRAPROLIN EXPRESSION IN LESIONAL SKIN OF PATIENTS WITH NON SEGMENTAL VITILIGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, marwa khaled mahmoud, Resident AT DERMATOLOGY department-sohag hospital university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-07-11MS
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Non-segmental Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-segmental vitiligo (Active Comparator): patients with non-segmental vitiligo
  Interventions: Diagnostic Test: skin biopsy
- control group (Active Comparator)
  Interventions: Diagnostic Test: skin biopsy

INTERVENTIONS:
Diagnostic Test: skin biopsy — skin biopsy for immunohistochemical staining and assessment of tissue expression of tristetraprolin

SUMMARY:
Vitiligo is characterized by the selective loss of melanocytes, which in turn leads to totally amelanotic, non-scaly, chalky-white macule with distinct margins Vitiligo is the most common depigmenting skin disorder, with an estimated prevalence of 0.5-2% of the population in both adults and children worldwide Tumor necrosis factor (TNF-α), a pro-inflammatory cytokine is necessary for Th1 mediated response and immune homeostasis and the up-regulation of TNF-α can result in chronic inflammatory and autoimmune diseases . previous studies revealed a rise in transcript and protein levels of TNF-α in vitiligo patients The prime location of melanocytes, keratinocytes and fibroblasts is the epidermal microenvironment and these cells are capable of TNF-α expression and secretion TNF-α acts as an autocrine as well as a paracrine manner to suppress the melanocyte growth and proliferation ( Tristetraprolin (TTP) zinc finger protein 36 (ZFP36) is Ribonucleic acid (RNA) binding protein that preferentially binds to Adenylate-uridylate-rich (AU-rich) regions in the 3' untranslated regions (3'UTR) of target genes . Additionally, Tristetraprolin functions by destabilizing mRNAs encoding for oncogenes, cytokines (as TNFα), and chemokines involved in the inflammatory processes, by favoring their degradation and/or preventing their efficient translation The expression of proinflammatory mediator genes is tightly controlled by post-transcriptional regulation, which is mediated by a set of immune-related RNA binding proteins, such as tristetraprolin, Roquin, and Regnase

ELIGIBILITY:
Inclusion Criteria:

* This study will include adult patients>18 yrs with non -segmental vitiligo attending the dermatology outpatient clinics at Sohag University, Egypt. A group of participants will be included as a control group.This control group will be taken from patients seeking for abdominoplasty in plastic surgery department at Sohag University Hospital.

Exclusion Criteria:

- 1)Pregnancy. 2)Patients with chronic inflammatory skin disorders. 3)Patients on antioxidants or anti-inflammatory drugs. 4)Patients on topical or systemic treatment for vitiligo in the last 4 weeks prior to enrollment in the study.

5)Patients with other autoimmune diseases as thyroiditis. lupus erythematosus and rheumatoid arthritis 6)Patients with diabetes mellitus (DM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
tristetraprolin | 12 months
  Tristetraprolin (TTP) zinc finger protein 36 (ZFP36) is Ribonucleic acid (RNA) binding protein that preferentially binds to Adenylate-uridylate-rich (AU-rich) regions in the 3' untranslated regions (3'UTR) of target genes (Brooks et al., 2013). Additionally, Tristetraprolin functions by destabilizing mRNAs encoding for oncogenes, cytokines (as TNFα), and chemokines involved in the inflammatory processes, by favoring their degradation and/or preventing their efficient translation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alghamdi KM, Khurrum H, Taieb A, Ezzedine K. Treatment of generalized vitiligo with anti-TNF-alpha Agents. J Drugs Dermatol. 2012 Apr;11(4):534-9. PMID 22453596
- [Background] Alikhan A, Felsten LM, Daly M, Petronic-Rosic V. Vitiligo: a comprehensive overview Part I. Introduction, epidemiology, quality of life, diagnosis, differential diagnosis, associations, histopathology, etiology, and work-up. J Am Acad Dermatol. 2011 Sep;65(3):473-491. doi: 10.1016/j.jaad.2010.11.061. PMID 21839315
- [Background] Alkhateeb A, Fain PR, Thody A, Bennett DC, Spritz RA. Epidemiology of vitiligo and associated autoimmune diseases in Caucasian probands and their families. Pigment Cell Res. 2003 Jun;16(3):208-14. doi: 10.1034/j.1600-0749.2003.00032.x. PMID 12753387
- [Background] Brooks SA, Blackshear PJ. Tristetraprolin (TTP): interactions with mRNA and proteins, and current thoughts on mechanisms of action. Biochim Biophys Acta. 2013 Jun-Jul;1829(6-7):666-79. doi: 10.1016/j.bbagrm.2013.02.003. Epub 2013 Feb 18. PMID 23428348